CLINICAL TRIAL: NCT02178358
Title: A Randomized Phase 2 Study of LY2157299 Versus LY2157299 - Sorafenib Combination Versus Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of LY2157299 in Participants With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15065; H9H-MC-JBAS (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-06-12; First posted 2014-06-30 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: transforming growth factor beta (TGF-β)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Camurati-Engelmann Syndrome | interventions — LY-2157299; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 150 milligram (mg) Galunisertib Monotherapy (Experimental): 150 mg galunisertib administered orally, twice daily (BID) for 14 days followed by 14 days with no study drug (28 days cycle).
  Interventions: Drug: LY2157299
- 150 mg Galunisertib + 400 mg Sorafenib Therapy (Experimental): 150 mg galunisertib administered orally, BID for 14 days followed by 14 days with no study drug (28 days cycle).
  400 mg sorafenib administered orally BID for 28 days.
  Interventions: Drug: LY2157299; Drug: Sorafenib
- 400 mg Sorafenib + Placebo Therapy (Placebo Comparator): Placebo administered orally BID for 14 days followed by 14 days with no study drug (28 days cycle).
  400 mg sorafenib administered orally BID for 28 days.
  Interventions: Drug: Sorafenib; Drug: Placebo

INTERVENTIONS:
Drug: LY2157299 — Administered orally
  Arms: 150 mg Galunisertib + 400 mg Sorafenib Therapy; 150 milligram (mg) Galunisertib Monotherapy
Drug: Sorafenib — Administered orally
  Arms: 150 mg Galunisertib + 400 mg Sorafenib Therapy; 400 mg Sorafenib + Placebo Therapy
Drug: Placebo — Administered orally
  Arms: 400 mg Sorafenib + Placebo Therapy

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as LY2157299 in participants with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have histological evidence of a diagnosis of HCC not amenable to curative surgery.
* Have Child-Pugh Class A.
* Have the presence of measurable disease.
* Have adequate organ function.
* Have a performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* If male or female with reproductive potential, must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug.
* If females with childbearing potential, must have had a negative serum pregnancy test 7 days prior to the first dose of study drug.
* Are able to swallow capsules or tablets.
* Have available diagnostic or biopsy tumor tissue.

Exclusion Criteria:

* Have received previous systemic treatment for advanced disease.
* Have known HCC with fibro-lamellar or mixed histology.
* Have presence of clinically relevant ascites.
* Have had a liver transplant.
* Have moderate or severe cardiac disease.
* Have active or uncontrolled clinically serious hepatitis B virus or hepatitis C virus infection.
* Have experienced Grade 3 or 4 gastrointestinal bleeding or any variceal bleeding episode in the 3 months prior to enrollment requiring transfusion or endoscopic or operative intervention.
* Have esophageal or gastric varices that require immediate intervention or represent a high bleeding risk.
* Had major surgery within 4 weeks prior to the study randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- China (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bengbu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
- Hong Kong (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hong Kong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kowloon
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwei Shan Township
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liouying/Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puzih City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow, participants who completed were those who died due to any cause or were alive and on study at conclusion but off treatment.
Period: Overall Study
Arm/Group | 150 Milligram (mg) Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Started | 20 | 74 | 38
Received at Least 1 Dose of Study Drug | 20 | 74 | 38
Completed | 19 | 72 | 36
Not Completed | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 150 mg Galunisertib Monotherapy: 150 mg galunisertib administered orally, BID for 14 days followed by 14 days with no study drug (28 days cycle).
- Total: Total of all reporting groups
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy | Total
Number analyzed (Participants) | 20 | 74 | 38 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 55 | 28 | 96
  >=65 years | 7 | 19 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.8) | 59.0 (8.5) | 58.6 (11.8) | 59.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 1 | 17
  Male | 16 | 62 | 37 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 74 | 38 | 132
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 7 | 33 | 13 | 53
  Hong Kong | 6 | 10 | 6 | 22
  China | 0 | 15 | 8 | 23
  Taiwan | 7 | 11 | 9 | 27
  Thailand | 0 | 5 | 2 | 7
Weight [Median (Full Range); unit: kilogram (kg)] | 66.400 [40.00 to 83.20] | 63.575 [39.70 to 87.00] | 62.400 [51.10 to 82.15] | 63.575 [39.70 to 87.00]
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 162.84 (7.38) | 165.30 (7.50) | 166.55 (5.69) | 165.29 (7.05)
BMI [Mean (Standard Deviation); unit: kilogram per square metre (kg/m2)] | 24.806 (4.105) | 23.224 (3.248) | 22.843 (3.062) | 23.354 (3.373)
Tobacco use [Count of Participants; unit: Participants]
  Never | 7 | 28 | 11 | 46
  Former | 7 | 35 | 22 | 64
  Current | 6 | 11 | 5 | 22
Alcohol use [Count of Participants; unit: Participants]
  Never | 7 | 29 | 16 | 52
  Former | 0 | 1 | 2 | 3
  Current | 13 | 44 | 20 | 77
Alcohol drinks per week [Mean (Standard Deviation); unit: Standard alcohol drinks per week] | 5.7 (7.2) | 3.3 (4.7) | 2.3 (2.8) | 3.4 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS): Number of Events
Description: OS defined as the time from the date of randomization to the date of death due to any cause. An overall survival event was defined as death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive. The number of participants with overall survival events (deaths) is reported.
Time Frame: Randomization to Date of Death from Any Cause (Up To 24 Months)
Population: All randomized participants. Censored participants: Galunisertib Monotherapy =5, Galunisertib Plus Sorafenib Therapy = 16 and Sorafenib Plus Placebo Therapy = 7.
Measure: Number; unit: Participants with events
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 20 | 74 | 38
Participants with events | 15 | 58 | 31
Statistical Analysis 1: Comparison: 150 mg Galunisertib Monotherapy vs 400 mg Sorafenib + Placebo Therapy; Test type: Superiority; p = 0.837, Bayesian exponential-likelihood model; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.434 to 1.226]
Statistical Analysis 2: Comparison: 150 mg Galunisertib + 400 mg Sorafenib Therapy vs 400 mg Sorafenib + Placebo Therapy; Test type: Superiority; p = 0.704, Bayesian exponential-likelihood model; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.633 to 1.266]

2. Secondary Outcome: Population Pharmacokinetics (PopPK): Mean Population Clearance of Galunisertib
Description: Population mean (between-subject coefficient variance [CV %]) apparent clearance.
Time Frame: Cycle (C) 1: Day (D)1: Predose, 0.5-2 hours(h) Postdose; D14: Predose, 0.5-2, 3-5 h, Postdose; D15 Morning; D22 Morning; Predose C2 and C3 Predose D1
Population: All randomized participants who received at least one dose of study drug, with evaluable galunisertib PK data. The analyses conducted on galunisertib exposure parameter from both arms combined per the statistical analysis plan, as monotherapy and combination arm showed no difference in galunisertib PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Groups:
- Galunisertib Monotherapy and Galunisertib + Sorafenib Therapy: 150 mg galunisertib administered orally, BID for 14 days followed by 14 days with no study drug (28 days cycle).
  150 mg galunisertib administered orally, BID for 14 days followed by 14 days with no study drug (28 days cycle). 400 mg sorafenib administered orally BID for 28 days.
Arm/Group | Galunisertib Monotherapy and Galunisertib + Sorafenib Therapy
Number analyzed (Participants) | 91
Liter per hour (L/hr) | 33.6 (48)

3. Secondary Outcome: Population Pharmacokinetics (PopPK): Steady State Apparent Volume of Distribution (Vss) of Galunisertib
Description: Population Vss [distribution of galunisertib in the body at steady state] after a single dose of galunisertib.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Galunisertib Monotherapy and Galunisertib + Sorafenib Therapy
Number analyzed (Participants) | 91
Liters (L) | 192 (69)

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP at initial treatment was defined as the number of months between date of randomization and the date of first documented disease progression or the date of death due to disease under study, whichever came first. Progression was assessed by the Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.Progressive Disease (PD)is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Randomization to the Date of Objective Progressive Disease or Date of Death due to Study Disease, whichever came first (Up To 24 Months)
Population: All randomized participants. Censored participants: Galunisertib Monotherapy =2, Galunisertib Plus Sorafenib Therapy = 15 and Sorafenib Plus Placebo Therapy = 9.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 20 | 74 | 38
Months | 1.41 [1.38 to 2.76] | 2.86 [2.63 to 4.21] | 4.14 [2.76 to 8.21]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Randomization to Measured Progressive Disease or Death (Up To 24 Months)
Population: All randomized participants. Censored participants: Galunisertib Monotherapy =1, Galunisertib Plus Sorafenib Therapy = 8 and Sorafenib Plus Placebo Therapy = 5.
Measure: Median (99% Confidence Interval); unit: Months
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 20 | 74 | 38
Months | 1.41 [1.38 to 2.76] | 2.86 [2.63 to 4.07] | 4.14 [2.76 to 5.59]

6. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Randomization to Measured Progressive Disease (Up To 24 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 20 | 74 | 38
Percentage of participants | 0.05 [0.001 to 0.249] | 0.027 [0.003 to 0.094] | 0.158 [0.060 to 0.313]

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Score
Description: EORTC QLQ-C30 consists of 30 items covered by 1 of 3 dimensions:
  1. Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  2. Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  3. Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
Time Frame: Baseline, 24 Months
Population: All randomized participants who received at least one dose of study drug and with baseline and post-baseline EORTC QLQ-C30 data for each EORTC QLQ-C30 items.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 19 | 65 | 35
units on a scale
  Global health status | 43.42 (23.171) | 55.90 (22.473) | 58.57 (17.326)
  Functional scale: Physical functioning | 84.56 (16.338) | 82.87 (19.613) | 80.95 (16.580)
  Functional scale: Role functioning | 89.47 (14.918) | 82.05 (24.880) | 85.24 (19.289)
  Functional Scale: Emotional Functioning | 84.65 (18.271) | 87.18 (17.247) | 86.90 (13.898)
  Functional Scale: Cognitive Functioning | 89.47 (16.860) | 91.03 (14.754) | 85.71 (18.142)
  Functional Scale: Social Functioning | 83.33 (24.845) | 84.10 (19.859) | 84.29 (18.052)
  Symptom Scale: Fatigue | 21.05 (23.393) | 24.10 (22.444) | 25.40 (18.390)
  Symptom Scale: Nausea and Vomiting | 2.63 (8.358) | 3.85 (8.725) | 3.33 (8.856)
  Symptom scale: Pain | 17.54 (19.621) | 17.18 (25.340) | 14.76 (20.521)
  Symptom scale: Dyspnoea | 17.54 (28.040) | 11.79 (19.922) | 12.38 (18.232)
  Symptom scale: Insomnia | 21.05 (31.838) | 9.74 (19.296) | 16.19 (16.903)
  Symptom scale: Appetite loss | 15.79 (25.744) | 16.92 (25.768) | 18.10 (23.351)
  Symptom scale: Constipation | 5.26 (12.488) | 6.15 (13.033) | 6.67 (15.760)
  Symptom scale: Diarrhoea | 10.53 (19.413) | 4.62 (13.013) | 10.48 (17.660)
  Symptom scale: Financial difficulties | 15.79 (25.744) | 23.08 (26.954) | 20.95 (22.989)

8. Secondary Outcome: Change From Baseline in EORTC QLQ Hepatocellular Carcinoma (HCC-18) Questionnaire Score
Description: The EORTC QLQ-HCC-18 was an 18-item questionnaire design used along with the 30-item EORTC QLQ-C30. EORTC QLQ-HCC 18 questionnaire included 8 symptom scales such as abdominal swelling, sex life, fatigue, body image, jaundice, nutrition, pain and fever. Each individual item ranges from 1 to 4, where 1 = "not at all" and 4 = "very much." All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a symptom scale/item represented a high level of symptomatology/problem.
Time Frame: Baseline, 24 Months
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC-QLQ HCC-18 data for each EORTC-QLQ HCC-18 items.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
Number analyzed (Participants) | 19 | 65 | 35
units on a scale
  Abdominal swelling | 24.56 (33.040) | 32.82 (31.453) | 27.62 (24.899)
  Sex Life | 28.07 (31.940) | 58.97 (35.242) | 46.08 (35.783)
  Fatigue | 32.16 (21.563) | 47.86 (29.128) | 46.98 (26.278)
  Body Image | 28.07 (26.089) | 36.15 (22.930) | 31.90 (20.758)
  Jaundice | 20.18 (25.202) | 27.69 (25.392) | 25.24 (21.531)
  Nutrition | 22.46 (21.223) | 34.05 (23.456) | 34.48 (18.611)
  Pain | 25.44 (18.732) | 25.38 (21.471) | 30.95 (21.822)
  Fever | 14.04 (16.909) | 25.38 (25.019) | 20.48 (20.646)

ADVERSE EVENTS:
Time Frame: Up To 63 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 150 mg Galunisertib Monotherapy | 150 mg Galunisertib + 400 mg Sorafenib Therapy | 400 mg Sorafenib + Placebo Therapy
All-Cause Mortality (participants affected / at risk) | 15/20 | 58/74 | 31/38
Serious Adverse Events (participants affected / at risk) | 6/20 | 31/74 | 11/38
Other Adverse Events (participants affected / at risk) | 17/20 | 73/74 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg Galunisertib Monotherapy (N=20) | 150 mg Galunisertib + 400 mg Sorafenib Therapy (N=74) | 400 mg Sorafenib + Placebo Therapy (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (6) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 150 mg Galunisertib Monotherapy (N=20) | 150 mg Galunisertib + 400 mg Sorafenib Therapy (N=74) | 400 mg Sorafenib + Placebo Therapy (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 17 (26) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 8 (10) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 16 (18) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6)
Ascites (Gastrointestinal disorders) | 3 (3) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (3) | 10 (11) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 29 (51) | 22 (50)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 7 (9) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 14 (15) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 7 (10) | 10 (13)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 15 (19) | 4 (8)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (8) | 23 (28) | 14 (16)
Influenza like illness (General disorders) | 2 (3) | 7 (8) | 1 (2)
Malaise (General disorders) | 0 (0) | 4 (6) | 3 (4)
Mucosal inflammation (General disorders) | 0 (0) | 4 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 4 (4) | 6 (6)
Pain (General disorders) | 1 (1) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 1 (3) | 26 (43) | 5 (5)
Rash pustular (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (6)
Alanine aminotransferase increased (Investigations) | 2 (2) | 23 (40) | 15 (24)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 26 (42) | 15 (25)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 10 (12) | 3 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 11 (15) | 15 (22)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 5 (8) | 3 (9)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 8 (12) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 9 (9) | 5 (7)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (5)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 9 (14) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 19 (35) | 13 (21)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 5 (6) | 6 (6)
White blood cell count decreased (Investigations) | 0 (0) | 4 (6) | 5 (10)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 27 (28) | 12 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 9 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 10 (16) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 7 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 33 (74) | 13 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 4 (7)
Headache (Nervous system disorders) | 3 (3) | 7 (8) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (6) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 7 (10) | 6 (9)
Genital disorder female (Reproductive system and breast disorders) | 0/4 (0) | 1/12 (1) | 0/1 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (9) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 15 (15) | 7 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (18) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (5) | 42 (57) | 19 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 13 (20) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 20 (24) | 9 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (11) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 15 (15) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of less than 90 days from the time submitted to the sponsor for review.The PI will remove from publication the information which the sponsor reasonably thinks would jeopardize its intellectual property interests or delay the publication until the publication no longer jeopardizes its intellectual property interests.

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT02178358/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT02178358/SAP_001.pdf